CLINICAL TRIAL: NCT02168309
Title: Comparison of Oral Nifedipine to Oral Labetolol for the Management of Severe Postpartum Hypertension
Brief Title: Oral Nifedipine Versus Oral Labetalol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Kilpatrick, Chair, Department of Obstetrics & Gynecology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro34034
Record Dates: First submitted 2014-06-17; First posted 2014-06-20 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Severe Postpartum Hypertension
MeSH Terms: interventions — Labetalol; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Labetalol (Other): Labetalol 200mg PO BID starting dose
  Interventions: Drug: Labetalol
- Nifedipine (Other): Nifedpine XL starting at dose 30mg PO daily
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Labetalol — Titrate up for blood pressure control
  Other Names: Oral labetalol starting at dose 200mg PO BID
  Arms: Labetalol
Drug: Nifedipine — Titrate up to achieve blood pressure control
  Other Names: Oral nifedipine 30mg XL PO starting
  Arms: Nifedipine

SUMMARY:
This study's aim is to determine whether oral extended release nifedipine is superior to oral labetolol for the management of postpartum severe hypertension, specifically time to achieve goal blood pressure, and shortening hospital stay. Our hypothesis is that oral extended release nifedipine is superior to oral labetolol for achieving goal blood pressure in the postpartum period.

DETAILED DESCRIPTION:
Hypertension complicating pregnancy is common and, when uncontrolled, can have devastating consequences. While the true incidence of postpartum hypertension is unknown, blood pressure (BP) is known to initially decrease 48 hours following delivery then peak on postpartum days 3-6, likely 45 from the mobilization of interstitial fluids following parturition.

The American College of Obstetricians and Gynecologists (ACOG) recommends medical treatment of persistent postpartum hypertension, defined as systolic BP (SBP) ≥150 mmHg or diastolic BP (DBP) ≥100 mmHg, on two or more occasions 4-6 hours apart. Prior studies compared intravenous medications to intramuscular and immediate-release oral 50 medications in the treatment of postpartum hypertension. However, oral labetalol and oral extended release nifedipine are the most commonly used medications for post- partum hypertension, and their efficacy has not been directly compared.

Our aim was to determine whether oral labetalol is associated with a shorter time to BP control compared to oral extended release nifedipine for management of persistent 55 postpartum hypertension. Our primary outcome was time to sustained BP control defined as the absence of severe hypertension (SBP ≥160 mmHg or DBP ≥105 mmHg) for at least 12 hours. Secondary outcomes included postpartum length of stay, need for increased dosing, need for additional oral antihypertensive agents, and patient-reported side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with the abililty to give informed consent
* Intrauterine pregnancy ≥ 32 weeks
* Postpartum
* Persistent postpartum blood pressures ≥ 160/105 on two or more occasions
* Primary obstetrician amenable to starting either study medication in the postpartum period

Exclusion Criteria:

* Use of other oral antihypertensives concomitantly
* Known AV heart block
* HR <60 or >120
* Absolute contraindication to nifedipine or labetolol such as allergy
* Significant renal disease (Cr >1.5 mg/dL)
* Heart failure
* Moderate persistent or severe asthma
* Preexisting diagnosis of chronic hypertension with medical treatment before delivery
* Chronic hypertension

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kilpatrick, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Sharma KJ, Greene N, Kilpatrick SJ. Oral labetalol compared to oral nifedipine for postpartum hypertension: A randomized controlled trial. Hypertens Pregnancy. 2017 Feb;36(1):44-47. doi: 10.1080/10641955.2016.1231317. Epub 2016 Oct 27. PMID 27786578

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Labetalol | Nifedipine
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Labetalol | Nifedipine | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (7.4) | 33.3 (6.4) | 33.7 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 17 | 16 | 33
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (4.1) | 33.0 (7.8) | 31.7 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Time (Hours) to Attain Sustained Blood Pressure Goal After Treatment Initiated With Antihypertensive Medication
Description: Primary outcome
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Labetalol | Nifedipine
Number analyzed (Participants) | 25 | 25
hours | 37.6 (32.5) | 38.2 (27.6)

2. Secondary Outcome: Total Length of Hospital Stay in Days
Description: Secondary outcome
Time Frame: 0-10 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Labetalol | Nifedipine
Number analyzed (Participants) | 25 | 25
days | 4.0 (1.5) | 4.3 (2.3)

ADVERSE EVENTS:
Arm/Group | Labetalol | Nifedipine
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No